CLINICAL TRIAL: NCT02885389
Title: Molecular Characterization of a Cohort of 73 Patients With Infantile Spasms Syndrome
Brief Title: Molecular Genetics in Infantile Spasms
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2010.614
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Infantile Spasms; West Syndrome
Keywords: Infantile spasms; West syndrome; variant; mutation; CNV; sequencing
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Infantile Spasms syndrome (ISs) is a characterized by epileptic spasms occurring in clusters with an onset in the first year of life. West syndrome represents a subset of ISs that associates spasms in clusters, a hypsarrhythmia EEG pattern and a developmental arrest or regression. Aetiology of ISs is widely heterogeneous including many genetic causes. Many patients, however, remain without etiological diagnosis, which is critical for prognostic purpose and genetic counselling. In the present study, the investigators performed genetic screening of 73 patients with different types of ISs by array-CGH and molecular analysis of 5 genes: CDKL5, STXBP1, KCNQ2, and GRIN2A, whose mutations cause different types of epileptic encephalopathies, including ISs, as well as MAGI2, which was suggested to be related to a subset of ISs.

ELIGIBILITY:
Inclusion Criteria:

* Infantile spams or West syndrome

Exclusion Criteria:

* brain malformation
* clinical features of tuberous sclerosis
* abnormal metabolic assays

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infantile spams or West syndrome
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Presence of deleterious gene variants in candidate genes for infantile spasms/west syndrome and for deleterious Copy-Number variations (CNV). A pan-genome analysis by microarray | Day one